CLINICAL TRIAL: NCT02241278
Title: Preoperative Low-dose Ketamine Has no Preemptive Analgesic Effect in Opioid-naïve Patients Undergoing Colon Surgery When Nitrous Oxide is Used
Brief Title: Preoperative Ketamine Has no Preemptive Analgesic Effect in Patients Undergoing Colon Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Arquitecto Marcide (Other)
Collaborators: Complexo Hospitalario Universitario de A Coruña (Other)
Responsible Party: Principal Investigator, Beatriz Nistal Nuno, M.D., Complexo Hospitalario Universitario de A Coruña
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MK334037
Record Dates: First submitted 2014-09-11; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Pain, Postoperative
Keywords: colon surgery; ketamine; patient-controlled-analgesia; preemptive analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): In the operating room, the anesthesiologist administered 50 mL of 0.9% saline intravenously to patients in the control group 30 minutes before surgical incision.
- Ketamine (Experimental): In the operating room, the anesthesiologist administered 0.5 mg/kg of ketamine chlorhydrate in 50 mL of 0.9 % saline intravenously to patients in the ketamine group 30 minutes before surgical incision. (a single dose).
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — In the operating room, the anesthesiologist administered 0.5 mg/kg of ketamine chlorhydrate in 50 mL of 0.9 % saline intravenously to patients in the ketamine group 30 minutes before surgical incision (a single dose).
  Other Names: ketamine chlorhydrate
  Arms: Ketamine

SUMMARY:
The analgesic properties of ketamine are associated with its non-competitive antagonism of the N-methyl-D-aspartate receptor; these receptors exhibit an excitatory function on pain transmission and this binding seems to inhibit or reverse the central sensitization of pain. In the literature, the value of this anesthetic for preemptive analgesia in the control of postoperative pain is uncertain. The objective of this study was to ascertain whether preoperative low-dose ketamine reduces postoperative pain and morphine consumption in adults undergoing colon surgery.

In a double-blind, randomized trial, 48 patients were studied. Patients in the ketamine group received 0.5 mg/kg intravenous ketamine before surgical incision, while the control group received normal saline. The postoperative analgesia was achieved with a continuous infusion of morphine at 0.015 mg∙kgˉ¹∙hˉ¹ with the possibility of 0.02 mg/kg bolus every 10 min. Pain was assessed using the Visual Analog Scale (VAS), morphine consumption, and hemodynamic parameters at 0, 1, 2, 4, 8, 12, 16, and 24 hours postoperatively. We quantified times to rescue analgesic (Paracetamol), adverse effects and patient satisfaction.

DETAILED DESCRIPTION:
In spite of the techniques we have at our disposal and the elementary nature of incisional pain, optimal pain management remains a challenge. Because the severity of early postoperative pain relates to residual pain after some types of surgery, perioperative pain management can considerably influence the long-term quality of life in patients.

Woolf, in 1983, first introduced the theory of preemptive analgesia to attenuate postoperative pain, confirming the presence of a central factor of post-injury pain hypersensitivity in experimental research. After this, experimental studies showed that various anti-nociceptive methods applied before injuries were more effective in reducing post-injury central sensitization in contrast to administration after injury.

After activation of C-fibers by noxious stimuli, sensory neurons become more sensitive to peripheral inputs, a process called central sensitization. 'Wind up, another mechanism activating spinal sensory neurons, is seen after reiterated stimulation of C-fibers. These sensitizations produce c-fos expression in sensory neurons, and are related to the activation of N-methyl-D-aspartic acid (NMDA) and neurokinin receptors. These genes produce long-lasting changes in the pain-processing system, resulting in hyperexcitation. According to Wall, protection of sensory neurons against central sensitization may provide relief from pain after surgery. Based on this assumption, preemptive analgesia has been recommended as an effective aid to control postsurgical pain. NMDA antagonists have been demonstrated to block the induction of central sensitization and revoke the hypersensitivity once it is established.

Ketamine is an old drug that is increasingly being considered for the treatment of acute and chronic pain. Its pharmacology and mechanism of action as an NMDA receptor antagonist are adequately known, but in clinical practice it presents irregular results. Since ketamine is an NMDA-receptor antagonist, it is supposed to avoid or revoke central sensitization, and thus to attenuate postoperative pain.

This antihyperalgesic action can be achieved by smaller doses than those required for anesthesia. Small-dose ketamine has been specified as not more than 1 mg/kg when given as an iv bolus, and not higher than 20 µg∙kgˉ¹∙minˉ¹ when given as a constant infusion.

Low-doses preemptive ketamine administered iv seem to reduce postoperative pain and/or analgesic consumption. According to one study, a single dose of ketamine 1 mg/kg, when administered in conjunction with local anesthetics, opioids or other anesthetics, provides good postoperative pain control.

Regardless of the overwhelming effectiveness of preemptive ketamine in animal experiments, clinical reports are mixed; some authors have described positive effects while others have not.

While early reviews of clinical findings were mostly contradictory, there is still conviction in the effectiveness of preemptive analgesia.

To our knowledge, no prior controlled study has determined the effectiveness of preoperative low-dose iv ketamine as contrasted with placebo in adults after open colon surgery. Thus, this clinical trial was designed to examine the postoperative analgesic effectiveness and opioid-sparing effect of single low-dose iv ketamine in contrast with placebo administered preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* normal Body Mass Index (18.5 - 24.9)
* American Society of Anesthesiologists (ASA) class I, II or III
* elective surgery
* surgery time between 60-150 min
* understanding of the Visual Analog Scale (VAS)
* lack of allergies or intolerance to anesthetics
* absence of psychiatric illness

Exclusion Criteria:

* cognitive deterioration
* inability to use the Patient-Controlled-Analgesia (PCA) device
* history of chronic pain syndromes
* chronic use of analgesics, sedatives, opioids or steroids
* liver or hematologic disease,
* history of drug or alcohol abuse
* intolerance to ketamine or Paracetamol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2001-09; Primary Completion 2002-06 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) score | at 0 hours postoperatively (arrival at recovery room)
  The VAS represents a scale with the lowest value as 0 (no pain) and the highest value as 10 (worst imaginable pain).
Visual Analog Scale (VAS) score | at 1 hour postoperatively
  The VAS represents a scale with the lowest value as 0 (no pain) and the highest value as 10 (worst imaginable pain).
Visual Analog Scale (VAS) score | at 2 hours postoperatively
  The VAS represents a scale with the lowest value as 0 (no pain) and the highest value as 10 (worst imaginable pain).
Visual Analog Scale (VAS) score | at 4 hours postoperatively
  The VAS represents a scale with the lowest value as 0 (no pain) and the highest value as 10 (worst imaginable pain).
Visual Analog Scale (VAS) score | at 8 hours postoperatively
  The VAS represents a scale with the lowest value as 0 (no pain) and the highest value as 10 (worst imaginable pain).
Visual Analog Scale (VAS) score | at 12 hours postoperatively
  The VAS represents a scale with the lowest value as 0 (no pain) and the highest value as 10 (worst imaginable pain).
Visual Analog Scale (VAS) score | at 16 hours postoperatively
  The VAS represents a scale with the lowest value as 0 (no pain) and the highest value as 10 (worst imaginable pain).
Visual Analog Scale (VAS) score | at 24 hours postoperatively
  The VAS represents a scale with the lowest value as 0 (no pain) and the highest value as 10 (worst imaginable pain).

SECONDARY OUTCOMES:
morphine consumption | at 0, 1, 2, 4, 8, 12, 16, and 24 hours postoperatively
  The cumulative amounts of morphine (mg) administered through the Patient-Controlled-Analgesia (PCA) device as a basal infusion and the incremental supplemental bolus required by the patient were documented at these time points.

OTHER OUTCOMES:
Blood Pressure (BP) systolic | at 0, 1, 2, 4, 8, 12, 16, and 24 hours postoperatively
  Measured in mm Hg. We evaluated these hemodynamic parameters as an indirect measure of pain.
Blood Pressure (BP) diastolic | at 0, 1, 2, 4, 8, 12, 16, and 24 hours postoperatively
  Measured in mm Hg. We evaluated these hemodynamic parameters as an indirect measure of pain
Heart rate | at 0, 1, 2, 4, 8, 12, 16, and 24 hours postoperatively.
  We evaluated these hemodynamic parameters as an indirect measure of pain
Respiratory rate | at 0, 1, 2, 4, 8, 12, 16, and 24 hours postoperatively.
  We evaluated these hemodynamic parameters as an indirect measure of pain.
Time for the first demand of analgesia | 24 h postoperatively.
  The time interval to first solicited rescue analgesia in the 24 h postoperatively (in minutes). This rescue analgesia was administered if the established analgesic treatment was not sufficient to alleviate pain.
Number of rescue doses | 24 h postoperatively
  The number of times a rescue analgesic dose was administered as a supplement in the first postoperative 24 hours.
Satisfaction score | 24 hours postoperatively
  Global patient satisfaction (0-3), regarding pain control, was measured 24 hours after the operation
Side effects | 24 hours postoperatively
  Number of Participants with Serious and Non-Serious Adverse Events in the 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Camba Rodriguez, M.D., Study Chair — Hospital Arquitecto Marcide; Beatriz Nistal Nuno, M.D., Principal Investigator — Complexo Hospitalario Universitario A Coruna; Enrique Freire-Vila, M.D., Study Director — Complexo Hospitalario Universitario A Coruna; Francisco Castro Seoane, M.D., Principal Investigator — Hospital Arquitecto Marcide
Locations (1):
- Hospital Arquitecto Marcide, Ferrol, A Coruna, Spain